CLINICAL TRIAL: NCT00124189
Title: A Phase I, Sequential Cohort, Dose Escalation Trial to Determine the Safety, Tolerability, and Maximum Tolerated Dose of GRN163L in Patients With Chronic Lymphoproliferative Disease
Brief Title: Safety and Dose Study of GRN163L to Treat Patients With Chronic Lymphoproliferative Disease(CLD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Geron Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GRN163L CP04-151
Record Dates: First submitted 2005-07-25; First posted 2005-07-27 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Chronic Lymphoproliferative Diseases
Keywords: Chronic lymphocytic leukemia; T-cell prolymphocytic leukemia; Chronic lymphoproliferative diseases; Telomerase; Telomerase Inhibition
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Prolymphocytic, T-Cell | interventions — GRN163L peptide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- open label (Other): Sequential dose cohort, open label, escalation trial evaluating one infusion duration of 2 hours
  Interventions: Drug: GRN163L

INTERVENTIONS:
Drug: GRN163L — Weekly intravenous infusion

SUMMARY:
The purpose of this study is to determine the safety and maximum tolerated dose of GRN163L in treating patients with refractory or relapsed chronic lymphoproliferative disease.

DETAILED DESCRIPTION:
Imetelstat Sodium (GRN163L) is a telomerase template antagonist with in vitro and in vivo activity in a variety of tumor model systems. Telomerase is an enzyme that is active primarily in tumor cells and is crucial for the indefinite growth of tumor cells. Inhibition of telomerase may result in antineoplastic effects. High telomerase levels and short telomere lengths correlate with other markers of poor prognosis in patients with chronic lymphoproliferative disease.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Male or female
* Chronic lymphoproliferative disease with related biology or similar clinical pattern to B-Cell Leukemia (CLL)including: small lymphocytic lymphoma (SLL), T cell prolymophocytic leukemia (T-PLL), B cell prolymphocytic leukemia (B-PLL), mantle cell lymphoma or other non-Hodgkins lymphoma in leukemic phase (peripheral blood circulating malignant cells present), Waldenstrom's macroglobulinemia
* Must have relapsed from or be refractory to prior therapeutic regimens
* Patients with CLL or SLL must have received at least one prior purine analogue-based chemotherapy regimen (eg, fludarabine, pentostatin or cladribine)
* If previously treated with an anthracycline, anthracenedione, or trastuzumab, must have left ventricular ejection fraction > 50%
* ECOG performance status 0-2
* Life expectancy 3 months or greater

Exclusion Criteria:

* Pregnant or lactating women
* Active 2nd malignancy or history of another malignancy within 2 years, except:treated, non-melanoma skin cancer,treated breast or cervical carcinoma in situ,or resected T1a or b prostate cancer
* Chemotherapeutic agents within 4 weeks prior to study
* High dose CTX with stem cell support within 6 months prior to study
* Signal transduction inhibitors,or monoclonal antibodies within 4 weeks prior to study
* Immunotherapy or biological response modifiers within 4 weeks prior to study
* Systemic hormonal therapy within 4 weeks prior to study
* Anticoagulant therapy, antiplatelet therapy within 2 weeks prior to study
* Radiotherapy within 4 weeks prior to study
* Active autoimmune disorder
* Central nervous system or leptomeningeal involvement
* Clinically significant cardiovascular disease
* Known HIV infection
* Serious/active infection
* Surgical procedure within 2 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2005-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Safety, tolerability, dose-limiting toxicities (DLT), and maximum tolerated dose (MTD) or recommended phase II dose of GRN163L in patients with relapsed or refractory chronic lymphoproliferative disease | First 3 weeks

SECONDARY OUTCOMES:
PK and PD | Measured in the first 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Kelsey, MD, Study Director — Geron Corporation
Locations (8):
- United States (8):
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Center, Buffalo, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Weill Medical College of Cornell University, New York, New York
  - The Ohio State University James Cancer Hospital, Columbus, Ohio
  - UT Southwestern, Dallas, Texas
  - University of Texas Health Science Center, San Antonio, Texas

REFERENCES:
- See also: Sponsor company web page. — http://www.geron.com